CLINICAL TRIAL: NCT01642381
Title: Component Analysis for Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Morgenstern, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA 020077-01A1
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Alcohol-Related Disorders; Alcohol Use Disorders; Alcohol Drinking; Alcoholism; Alcohol Abuse
Keywords: Drinking; Alcohol Problems; Alcoholism; Moderation-Oriented Treatment; Controlled Drinking; Reduced Drinking; Heavy Drinking; Problematic Drinking; Non-Abstinence-based Drinking
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Alcohol Drinking | interventions — Receptor-Like Protein Tyrosine Phosphatases, Class 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychotherapy (Active Comparator)
  Interventions: Behavioral: Full Motivational Interviewing ("FMI"); Behavioral: Spirit Only Motivational Interviewing ("SOMI")
- Self-Change Control ("SCC") (No Intervention): SCC participants will be told that they should attempt to reduce their drinking over the course of 8 weeks. (If unsuccessful, they will be offered Full Motivational Interviewing therapy sessions.)

INTERVENTIONS:
Behavioral: Full Motivational Interviewing ("FMI") — Relational and technical technical (directive) strategies in counselling sessions to significantly increase commitment strength to reduce drinking.
  Arms: Psychotherapy
Behavioral: Spirit Only Motivational Interviewing ("SOMI") — Empathic and non-directive counselling based on Rogerian psychotherapy model.
  Arms: Psychotherapy

SUMMARY:
The purpose of this study is to investigate the critical components of motivational interviewing (MI), a psychotherapeutic intervention, in reducing heavy or problematic drinking. The study will disaggregate MI into its component parts and test full MI compared to MI without its directive strategies. This study will test whether the directive elements of MI are critical or whether MI effects may be attributable solely to its Rogerian, non-directive components. For more information, go to http://caspirnyc.org/p_motion.html

DETAILED DESCRIPTION:
Project Motion is a clinical research study for people seeking to reduce, but not stop their drinking. Individuals who qualify will receive a comprehensive assessment and brief individual psychotherapy at no cost. The study is being conducted by a team of scientists at Columbia University College of Physicians and Surgeons and the New York State Psychiatric Institute and is funded by the National Institutes of Health (NIH). Our offices are located next to Columbus Circle and we offer convenient hours for appointments.

The purpose of our study is to understand how brief psychotherapy helps people reduce alcohol consumption and drinking problems. For example, we know that some people can reduce drinking with little or no treatment, whereas others benefit from one-on-one psychotherapy. However, we do not know why this happens. Individuals who qualify and decide to participate will be assigned by chance to one of three conditions. Individuals assigned to the first two conditions will receive brief psychotherapy, beginning the first week of their participation in the study. Individuals in the third condition will receive feedback on their drinking and be asked to reduce their drinking with the aid of telephone self-monitoring for a period of 8 weeks. Individuals in the third condition will then receive psychotherapy as well. The delay of 8 weeks will allow us to understand how the psychotherapy works compared to how people change without counseling.

ELIGIBILITY:
Inclusion Criteria:

* Primary current diagnosis of Alcohol Use Disorder
* Meets DSM-IV criteria for inability to control or cut down on drinking
* Have an average weekly consumption of >24 standard drinks for men and >15 standard drinks for women
* Show no evidence of significant cognitive impairment
* Are willing to reduce drinking to non-hazardous levels
* Not seeking to quit drinking
* Agree not to seek additional substance abuse treatment during treatment period
* Fluent in English

Exclusion Criteria:

* Have a current DSM-IV diagnosis of drug dependence (other than nicotine/marijuana)
* Have a serious psychiatric illness (e.g., psychotic disorder, bipolar disorder, major depression) or substantial suicide or violence risk
* Have clinically severe alcoholism as evidenced by a history of significant medical problems associated with drinking, seizures or severe withdrawal symptoms, or an inpatient treatment episode for drinking
* Legally mandated to receive substance abuse treatment
* Sufficiently socially unstable as to preclude completion of study requirements (e.g., homeless)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-05; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back | 36 weeks
  Calendar-based method of recording drinking patterns. Data will be aggregated into summary variables including sum of standard drinks, mean drinks per drinking day, and percent days heavy drinking at multiple time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Morgenstern, PhD, Principal Investigator — North Shore LIJ Health Systems
Locations (1):
- North Shore LIJ Health Systems, Great Neck, New York, United States